CLINICAL TRIAL: NCT00637520
Title: Insulin Resistance in Nonalcoholic Fatty Liver Disease: A Case Control Study
Status: Terminated | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00006742; NIH K23 Award; 8592 (Other: Duke legacy protocol number)
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2016-09

CONDITIONS: Insulin Resistance; Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease; Insulin Resistance; Lipid Metabolism
MeSH Terms: conditions — Insulin Resistance; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen tissue, serum, whole blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Subjects with NAFLD
- 2: Subjects without liver disease
- 3: Subjects with non-steatotic hepatitis

SUMMARY:
We hypothesize that insulin resistance is characteristic of nonalcoholic fatty liver disease as compared to age, gender, non-diabetic BMI-matched control subjects, both healthy and those with non-cirrhotic, non-steatotic liver disease.

DETAILED DESCRIPTION:
Purpose of the study:

To date, no case control study evaluating insulin resistance (IR) in nonalcoholic fatty liver disease (NALFD) has been published. We hypothesize that IR is characteristic of NAFLD as compared to age, gender, non-diabetic BMI-matched control subjects, both healthy and those with non-cirrhotic, non-steatotic liver disease. The following aims test this central hypothesis:

Specific Aim 1: Measure IR and insulin clearance using intravenous glucose tolerance testing and Bergman's Minimal Modeling in patients with NAFLD as compared to matched controls (healthy and those with non-steatotic hepatitis). This aim tests the postulate that IR is necessary for the development of hepatic steatosis as compared to healthy (non-steatotic livers). It will also test the postulate that IR is not present as a confounding factor (impaired hepatic clearance) in NAFLD as compared to those with non-steatotic forms of hepatitis.

Specific Aim 2: Determine if IR is associated with altered parameters of lipid metabolism as compared to matched controls. This aim addresses whether IR (if present) is associated with abnormal lipid parameters in NAFLD or can be observed irrespective of the presence of hepatic steatosis.

Specific Aim 3: Measure the differential effects of IR and lipid metabolism on peripheral mononuclear cell (PBMC) inflammatory response and the associated hepatocyte mitochondrial ultrastructure and measures of oxidative stress. Since increased oxidative stress and bioenergetic failure have been associated with hepatic steatosis, this aim will address whether IR and/or steatosis results in impaired inflammatory response and increased oxidative stress as compared to controls. Changes in innate immune response will be determined by measuring inflammatory indices thought to correlate with obesity, IR, and/or chronic hepatitis: 1) interleukins (IL-2, IL-4, IL-6, IL-10, IL-12, IL-18) 2) C-reactive protein, 3) TNF-a and TGF-B 4) IFN-A & IFN-g, and 5) adiponectin. Changes in oxidative stress will be determined by measuring key indices of oxidative stress and damage. These include, a) reduced and oxidized glutathione (GSH and GSSG); oxidation/reduction status), b) malondialdehyde (MDA;lipid peroxidation), c) nitrotyrosine (NO damage), and d) 8OHdG and 8OHG (DNA damage).

Background and significance:

Obesity, diabetes, hypertriglyceridemia, hypertension, and coronary heart disease constitute a phenotype common to individuals with either the IR syndrome or NAFLD1-12. Furthermore, the hepatic steatosis, fibrosis, and cirrhosis characteristic of NAFLD are also frequent histologic findings in patients with IR 3-7. Together, these data beg the question whether NAFLD and IR are causally associated. Support for this notion derives from recent observations that IR may be a strong, independent predictor of NAFLD, even in the absence of glucose intolerance 13. Moreover, since NAFLD has been reported to occur in lean subjects (BMI greater than 25) with normoglycemia 14, 15, it is reasonable to postulate that NAFLD may be an early manifestation and a consequence of IR. Increased oxidative stress is an important pathogenic mechanism of obesity-associated metabolic syndrome 16. Fat accumulation correlated with systemic oxidative stress in humans and mice. However, increase oxidative stress as an instigator of the metabolic syndrome in patients with NAFLD as compared to controls has not yet been investigated. Furthermore, impaired cytokine medicated inflammatory response has been shown to correlate with body mass index across the broad range of obesity and may mediate hepatic steatosis and/or lead to mitochondrial dysfunction in hepatocytes 17, 18. Discerning whether NAFLD is attributable to increased oxidative stress and/or abnormalities in innate immune response would be imperative in identifying potentially useful therapeutic targets for obesity-associated liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Biochemical and liver histologic features to confirm the presence of a healthy liver, fatty liver, and/or non-fatty liver with inflammation due to another etiology besides NAFLD.

Exclusion Criteria:

* > 20 grams of alcohol/day
* Impaired oral glucose tolerance test
* Clinical or histologic evidence of cirrhosis (stage 5-6 fibrosis) or portal hypertension.
* Chronic hepatitis C infection
* Known diabetes mellitus or need for insulin-sensitizing agents and/or insulin therapy.
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Liver Clinic, Liver Transplant Clinic, Weight Loss Surgery Clinic
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2007-07; Primary Completion 2013-03-29 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
Measure Insulin Resistance (IR) and clearance its effects on lipid metabolism, inflammatory response, and oxidative stress using intravenous glucose tolerance testing in patients with NAFLD as compared to matched controls. | 36 months
Determine if IR is associated with altered parameters of lipid metabolism as compared to matched controls | 36 months
Measure the differential effects of IR and lipid metabolism on peripheral mononuclear cell (PBMC) inflammatory response and the associated hepatocyte mitochondrial ultrastructure and measures of oxidative stress. | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Manal F Abdelmalek, MD., MPH, Principal Investigator — Faculty Member
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Marchesini G, Brizi M, Morselli-Labate AM, Bianchi G, Bugianesi E, McCullough AJ, Forlani G, Melchionda N. Association of nonalcoholic fatty liver disease with insulin resistance. Am J Med. 1999 Nov;107(5):450-5. doi: 10.1016/s0002-9343(99)00271-5. PMID 10569299
- [Background] Ratziu V, Giral P, Charlotte F, Bruckert E, Thibault V, Theodorou I, Khalil L, Turpin G, Opolon P, Poynard T. Liver fibrosis in overweight patients. Gastroenterology. 2000 Jun;118(6):1117-23. doi: 10.1016/s0016-5085(00)70364-7. PMID 10833486
- [Background] Silverman JF, Pories WJ, Caro JF. Liver pathology in diabetes mellitus and morbid obesity. Clinical, pathological, and biochemical considerations. Pathol Annu. 1989;24 Pt 1:275-302. No abstract available. PMID 2654841
- [Background] Kern WH, Heger AH, Payne JH, DeWind LT. Fatty metamorphosis of the liver in morbid obesity. Arch Pathol. 1973 Nov;96(5):342-6. No abstract available. PMID 4741905
- [Background] Angulo P. Nonalcoholic fatty liver disease. N Engl J Med. 2002 Apr 18;346(16):1221-31. doi: 10.1056/NEJMra011775. No abstract available. PMID 11961152
- [Background] Chitturi S, Abeygunasekera S, Farrell GC, Holmes-Walker J, Hui JM, Fung C, Karim R, Lin R, Samarasinghe D, Liddle C, Weltman M, George J. NASH and insulin resistance: Insulin hypersecretion and specific association with the insulin resistance syndrome. Hepatology. 2002 Feb;35(2):373-9. doi: 10.1053/jhep.2002.30692. PMID 11826411
- [Background] Marchesini G, Bugianesi E, Forlani G, Cerrelli F, Lenzi M, Manini R, Natale S, Vanni E, Villanova N, Melchionda N, Rizzetto M. Nonalcoholic fatty liver, steatohepatitis, and the metabolic syndrome. Hepatology. 2003 Apr;37(4):917-23. doi: 10.1053/jhep.2003.50161. PMID 12668987
- [Background] Pagano G, Pacini G, Musso G, Gambino R, Mecca F, Depetris N, Cassader M, David E, Cavallo-Perin P, Rizzetto M. Nonalcoholic steatohepatitis, insulin resistance, and metabolic syndrome: further evidence for an etiologic association. Hepatology. 2002 Feb;35(2):367-72. doi: 10.1053/jhep.2002.30690. PMID 11826410
- [Background] Ikai E, Ishizaki M, Suzuki Y, Ishida M, Noborizaka Y, Yamada Y. Association between hepatic steatosis, insulin resistance and hyperinsulinaemia as related to hypertension in alcohol consumers and obese people. J Hum Hypertens. 1995 Feb;9(2):101-5. PMID 7752170
- [Background] DeFronzo RA, Ferrannini E. Insulin resistance. A multifaceted syndrome responsible for NIDDM, obesity, hypertension, dyslipidemia, and atherosclerotic cardiovascular disease. Diabetes Care. 1991 Mar;14(3):173-94. doi: 10.2337/diacare.14.3.173. PMID 2044434
- [Background] Marchesini G, Brizi M, Bianchi G, Tomassetti S, Bugianesi E, Lenzi M, McCullough AJ, Natale S, Forlani G, Melchionda N. Nonalcoholic fatty liver disease: a feature of the metabolic syndrome. Diabetes. 2001 Aug;50(8):1844-50. doi: 10.2337/diabetes.50.8.1844. PMID 11473047
- [Background] Bacon BR, Farahvash MJ, Janney CG, Neuschwander-Tetri BA. Nonalcoholic steatohepatitis: an expanded clinical entity. Gastroenterology. 1994 Oct;107(4):1103-9. doi: 10.1016/0016-5085(94)90235-6. PMID 7523217
- [Background] Lee JH, Rhee PL, Lee JK, Lee KT, Kim JJ, Koh KC, Paik SW, Rhee JC, Choi KW. Role of hyperinsulinemia and glucose intolerance in the pathogenesis of nonalcoholic fatty liver in patients with normal body weight. Korean J Intern Med. 1998 Feb;13(1):12-4. PMID 9538625
- [Background] Expert Committee on the Diagnosis and Clasification of Diabetes Mellitus. American Diabetes Association: clinical practice recommendations 2002. Diabetes Care. 2002 Jan;25 Suppl 1:S1-147. doi: 10.2337/diacare.25.2007.s1. No abstract available. PMID 11788484
- [Background] Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y, Nakayama O, Makishima M, Matsuda M, Shimomura I. Increased oxidative stress in obesity and its impact on metabolic syndrome. J Clin Invest. 2004 Dec;114(12):1752-61. doi: 10.1172/JCI21625. PMID 15599400
- [Background] Manes JL, Taylor HB, Starkloff GB. Relationship between hepatic morphology and clinical and biochemical findings in morbidly obese patients. J Clin Pathol. 1973 Oct;26(10):776-83. doi: 10.1136/jcp.26.10.776. PMID 4750460
- [Background] Kaneda M, Kashiwamura S, Ueda H, Sawada K, Sugihara A, Terada N, Kimura-Shimmyo A, Fukuda Y, Shimoyama T, Okamura H. Inflammatory liver steatosis caused by IL-12 and IL-18. J Interferon Cytokine Res. 2003 Mar;23(3):155-62. doi: 10.1089/107999003321532493. PMID 12716488
- [Background] Khaodhiar L, Ling PR, Blackburn GL, Bistrian BR. Serum levels of interleukin-6 and C-reactive protein correlate with body mass index across the broad range of obesity. JPEN J Parenter Enteral Nutr. 2004 Nov-Dec;28(6):410-5. doi: 10.1177/0148607104028006410. PMID 15568287